CLINICAL TRIAL: NCT07194317
Title: A Feasibility Study to Determine the Most Appropriate Digital Dietary Assessment Tool in Patients With Obesity Initiating GLP-1 Receptor Agonist Treatment
Acronym: FIDGET
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 347758
Record Dates: First submitted 2025-09-08; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Obese Patients
Keywords: Digital health; Diet Assessment; Acceptability testing

STUDY DESIGN:
Intervention Model Description: Over three weeks participants will be asked to record three consecutive days of dietary intake each week using a different tool. Participants will be assigned to an order they complete the three tools from six different sequence options. The order will be assigned based on auto number generation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Feasibility and acceptability (Other): Participants will record their dietary intake over three weeks, using a different tool for three consecutive days each week. The digital tools are: MyFood24, Nutritics-Libro and Intake24.The order sequence to complete will be from auto number generation.
  Interventions: Device: Testing 3 different digital dietary assessment tools in a random order (Nutritics-Libro, MyFood24 and Intake24)

INTERVENTIONS:
Device: Testing 3 different digital dietary assessment tools in a random order (Nutritics-Libro, MyFood24 and Intake24) — 55 participants will be recruited (target to complete the study n=50). The acceptability trial will be conducted remotely. A baseline questionnaire will capture demographic data. Over three weeks participants will be asked to record three random consecutive days of dietary intake each week using a different tool. Participants will be randomised to the order they complete the tools. To minimise potential biases. Participants will be randomly assigned to one of the six possible tool completion sequences (Table 1) using a relevant participant randomization package (e.g., rempsyc) in R (v4.4.2), which is a free, open-source statistical software used for data analysis and randomisation.

SUMMARY:
New medications that work on gut hormones such as semaglutide (Wegovy) and tirzepatide (Mounjaro) are helping many people lose weight and are now recommended for treating obesity by the NHS. While these treatments are effective for weight loss, we don't yet know how they affect what people eat or their overall nutrition. Understanding diet before, during, and after treatment is important. Traditional ways of tracking diet, like paper food diaries, can be difficult to use and are time consuming for clinicians to interpret and record in clinical notes. Digital tools like MyFood24, Nutritics-Libro, and Intake24 may offer a better way to record what people eat, but we need to find out if they can be easily used in everyday healthcare settings. The FIDGET study will test how well these digital diet tools can be used in clinics and linked with electronic health records. The study will use surveys and group discussions to understand how patients and healthcare professionals feel about using these tools.

DETAILED DESCRIPTION:
Gut hormone-based therapies including the glucagon-like peptide-1 (GLP-1) receptor agonist semaglutide (Wegovy) and dual glucose-dependent insulinotropic polypeptide (GIP)/ GLP-1 receptor agonist Tirzepatide (Mounjaro) are increasingly effective in weight management, leading to their recommendations for obesity treatment in the UK's National Health Service (NHS). These medications support weight loss; however, their impact on dietary intake and nutritional status remains unexplored. Assessing diet is essential before, during and after treatment. Several digital dietary assessment tools address limitations of traditional paper-based methods; however, feasibility of integrating these digital tools into routine clinical workflows has not been assessed. The Feasibility of Digital Dietary Assessment (FIDGET) study will evaluate integration of digital dietary recording tools (MyFood24, Nutritics-Libro and Intake24) into routine clinical workflows and electronic health record, using a randomised crossover design with mixed-methods evaluation (quantitative cross-sectional surveys, qualitative focus groups).

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >18 years
* Living with obesity as diagnosed by healthcare professional.
* Referral to T3WMS at GSTT and currently on the service waiting list
* Eligible for GLP-1 receptor agonist (Wegovy) prescription
* Have an active MyChart account
* Have an email address
* Access to a digital device such as a smart phone, computer or tablet where you can access the internet
* Not following a meal replacement diet, for example soups / shakes
* Able to provide informed consent.
* Able to complete surveys in English.

Exclusion Criteria:

* Adults aged >18 years

  * Living with obesity as diagnosed by healthcare professional.
  * Referral to T3WMS at GSTT and currently on the service waiting list
  * Eligible for GLP-1 receptor agonist (Wegovy) prescription
  * Have an active MyChart account
  * Have an email address
  * Access to a digital device such as a smart phone, computer or tablet where you can access the internet
  * Not following a meal replacement diet, for example soups / shakes
  * Able to provide informed consent.
  * Able to complete surveys in English.
  * Not able to provide informed consent
  * Not able to complete surveys in English
  * Has an eating disorder
  * Taking part in another research trial that involves dietary modification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Usability | Following each test period of 1 week
  Participants will complete a questionnaire to assess their experience and acceptability of using the tool. The System Usability Scale (SUS) will be used to measure the usability of the digital dietary assessment tools. A higher score denotes the system is more user friendly.
Usability and context of use | Following each test period of 1 week]
  Participants will complete a questionnaire to assess their experience and acceptability of using the tool. The modified version of the Rawl Usability Questionnaire - this measures the usability of specific features of digital applications and context of use.

SECONDARY OUTCOMES:
Patient experience and acceptability | Within 4 months of completion of the tool testing
  This is a qualitative outcome. A purposive sub-sample of 10 participants from the testing phase will be invited participate in one of two online focus groups to discuss their experiences of the dietary assessment tools. The focus group questions were designed to assess two main domains (patient experience and acceptability).The Quadruple Aim framework and the Theoretical Framework of Acceptability (TFA) guided the development of the questions to capture participants' overall experience including tool usability, perceived usefulness and accuracy, impact on daily routine and satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Guy's and St Thomas' NHS Trust, London, Southwark, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tanihara M, Suzuki Y, Yamamoto E, Noguchi A, Mizushima Y. Sustained release of basic fibroblast growth factor and angiogenesis in a novel covalently crosslinked gel of heparin and alginate. J Biomed Mater Res. 2001 Aug;56(2):216-21. doi: 10.1002/1097-4636(200108)56:23.0.co;2-n. PMID 11340591
- [Background] Polack FM. Modification of the immune graft response by azathioprine. Surv Ophthalmol. 1966 Aug;11(4):545-53. No abstract available. PMID 5331571
- [Background] Martin D. Postcodes and the 1991 census of population: issues, problems and prospects. Trans Inst Br Geogr. 1992;17(3):350-7. PMID 12157823
- [Background] van Eerde MR, Kampinga HH, Szabo BG, Vujaskovic Z. Comparison of three rat strains for development of radiation-induced lung injury after hemithoracic irradiation. Radiother Oncol. 2001 Mar;58(3):313-6. doi: 10.1016/s0167-8140(00)00301-7. PMID 11230893